CLINICAL TRIAL: NCT03378271
Title: Accuracy and Treatment Experience of Two Glucose Monitoring Systems Tested Simultaneously in Ambulatory Patients With Type 1 Diabetes and Renal Impairment
Brief Title: Accuracy and Treatment Experience of Two Glucose Monitoring Systems Tested in Patients With Type 1 Diabetes and Renal Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CGM renal impairment
Record Dates: First submitted 2017-12-11; First posted 2017-12-19 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus Complication; Renal Impairment
Keywords: Continuous Glucose Monitoring; Flash glucose Monitoring; Renal Impairment; Type 1 Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Complications; Renal Insufficiency; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FGM/CGM (Experimental): each patient will have a CGM and a FGM, subcutaneous glucose sensors, the data will be compared to the time-matched reference blood glucose measurements.
  Each ambulatory patient will sample capillary blood with the HemoCue meter and measure the concentration of glucose minimum 3 times per day for 14 days. The concentration of finger-stick capillary blood glucose will be measured using the self-monitoring blood glucose (SMBG) hemocue meter in their daily living. The subjects will record SMBG, in a written diary. Subjects will dose insulin according to their routine methods throughout the 14 day study
  Interventions: Device: Simultanious CGM/FGM

INTERVENTIONS:
Device: Simultanious CGM/FGM — Patients will use both CGM and FGM and document their values as well as documenting a capillary blood glucose value.

SUMMARY:
The study aims to evaluate the accuracy of two commercial glucose monitoring systems in patients with type 1 or type 2 diabetes and renal impairment, including patients with or without dialysis. Patients treatment experience will even be evaluated.

DETAILED DESCRIPTION:
Continuous glucose monitoring (CGM) and Flash glucose monitoring (FGM) are tools today mainly used in the treatment of patients with type 1 diabetes. Both glucose monitors are subcutaneous tissue sensors, which provide a tissue fluid glucose measurement every 1 to 5 minutes. The real-time glucose sensor trend data can help patients with diabetes better manage their insulin needs with meals and exercise. The following glucose monitoring systems are two of the most current sensor technologies available for clinical use the Dexcom G5 (Dexcom Corporation), and the FGM (Abbot Freestyle Libre).

High glucose levels in patients with type 1 or 2-diabetes lead to increased risks of micro- and macrovascular complications, while low glucose levels may lead to unconsciousness. Therefore, it is important for patients to manage glucose levels as close to normal (4-7 mmol/l) as possible. This is generally performed by appropriate dosage of different insulins, calculated from the preprandial glucose level, carbohydrate intake, and physical activity. In spite of careful dosage, glucose levels often become too low or too high.

CGM is a novel tool to detect low and high glucose levels, and it is capable of sounding an alarm for low and high glucose levels. CGM has been available in clinical practice in Sweden for approximately 5 years. FGM is as CGM also a novel tool to detect low and high glucose levels, but is not capable of sounding an alarm for low and high glucose levels. FGM has been available in clinical practice in Sweden since late 2014.

Since both CGM and FGM measure the glucose level by a sensor in subcutaneous tissue, there is uncertainty in the estimation of blood glucose levels. The accuracy of a certain CGM or FGM system can be assessed by comparing the glucose levels estimated by the glucose monitors with measured glucose levels in capillary blood samples. To our knowledge there are no studies comparing the accuracy of the Dexcom G5 sensor with the Freestyle Libre sensor. In the current study, we will compare the accuracy and treatment experience of these two glucose monitoring sensors available on the market for clinical use in patients with type 1 or 2 diabetes and renal impairment with an eGFR<30 ml/min both in and not in dialysis.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 or type 2 diabetes with renal impairment and eGFR <30 ml/min measured within the last three months.
2. Adult patients, age 18 or older and <80 years.
3. Written Informed Consent

Exclusion criteria:

1. Pregnancy
2. Patients with severe cognitive dysfunction or other disease which makes glucose monitoring use difficult.
3. Patients requiring continuous use of paracetamol. Paracetamol must not have been used the week before the study and shall not be used during the duration because it disturbs the interpretation of blood glucose levels estimated by the Dexcom G5. However, other pain killers can be used throughout the study period.
4. Current CGM or FGM use.
5. History of allergic reaction to any of the CGM or FGM materials or adhesives in contact with the skin.
6. History of allergic reaction to chlorhexidine or alcohol anti-septic solution.
7. Abnormal skin at the anticipated glucose sensor attachment sites (excessive hair, burn, inflammation, infection, rash, and/or tattoo).
8. Patients with renal impairment and eGFR greater or equal to 30 ml/min estimated by the MDRD formula.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-05-05 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Accuracy of CGM and FGM | The whole study period Day 1-14
  Evaluation of accuracy in estimating capillary glucose levels of two commercial glucose monitoring systems (CGM and FGM), Dexcom G5 system (Dexcom sensor) and the Abbot Freestyle Libre sensor, in ambulatory patients with type 1 or type 2 diabetes and renal impairment with an eGFR<30 ml/min both in and not in dialysis.

SECONDARY OUTCOMES:
The evaluation of the accuracy of the 2 glucose monitoring systems during each studied time interval (day 1-3 and day 4-6) | Day 1-6 of study period
  The evaluation of the accuracy of the 2 glucose monitoring systems for various glucose intervals (hypo, normo- and hyperglycaemia)
The evaluation of the accuracy of the 2 glucose monitoring systems for various glucose intervals (hypo, normo- and hyperglycaemia) | The whole study period Day 1-14
The evaluation of the accuracy of the 2 glucose monitoring systems during dialysis and not in dialysis | The whole study period Day 1-14
The evaluation of patients preferences and experience of the two glucose monitoring systems. | The whole study period Day 1-14
  Patients will answer questionnaires on both systems to see which system they prefer to use and find more user friendly. the questionnaire will be in the form of a Lickert scale from 0-10.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Lind, PhD, Principal Investigator — Gothenburgh University
Locations (1):
- NU-Hospital Group, Uddevalla, Sweden